CLINICAL TRIAL: NCT03925285
Title: Image Guided Surgery in Sinonasal Inverted Papilloma by Targeting Vascular Endothelial Growth Factor
Brief Title: Image Guided Surgery in Sinonasal Inverted Papilloma
Acronym: SNIPER
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. M.J.H. Witjes, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL66969.042.18
Record Dates: First submitted 2019-02-13; First posted 2019-04-24 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Inverted Papilloma; Molecular Fluorescence Imaging
MeSH Terms: conditions — Papilloma, Inverted

STUDY DESIGN:
Intervention Model Description: Patients are administered with bevacizumab-800CW. 2-4 days later, fluorescence imaging will be performed peroperatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV fluorescent tracer bevacizumab-800CW (Experimental): Patients will be administered with 10 or 25 bevacizumab-800CW.
  Interventions: Drug: Bevacizumab-800CW

INTERVENTIONS:
Drug: Bevacizumab-800CW — Two to four days prior to surgery bevacizumab-800CW will be administered intravenously
  Other Names: Bevacizumab-IRDye800CW

SUMMARY:
In sinonasal inverted papilloma (SNIP) it is very challenging to discriminate between tumor and surrounding tissue. Local recurrence is a frequent phenomenon as it occurs in 16.5% of the cases. There is need for an instrument that is able to guide the surgeon in removing all tumor tissue, whereas resection of healthy tissue is minimalized.

Molecular fluorescence guided surgery enables the visualization of targeted tumor-specific biomarkers by using fluorescence, thereby enhancing the contrast between normal mucosa and tumor tissue. The objective of this feasibility study is to determine if the intravenously administered conjugate bevacizumab-IRDye800CW accumulates more in SNIP than in normal sinonasal epithelium.

DETAILED DESCRIPTION:
Rationale: During surgical resection, it is very challenging to discriminate between sinonasal inverted papilloma (SNIP) and surrounding tissue, as SNIP is associated with inducement of granulomatous inflammation of the environment. As a result, the surgeon has to perform a thorough resection in order to remove the complete inverted papilloma, which is associated with substantial morbidity. Clearly, there is need for an instrument that is able to guide the surgeon to discriminate between SNIP and surrounding tissue. Molecular imaging techniques using targeted optical contrast agents is a promising technique to accommodate this need. Vascular Endothelial Growth Factor (VEGF) is overexpressed in SNIP compared to normal epithelium of the sinonasal area and has been used effectively in molecular imaging.

Objectives: The main objective is to study if the conjugate bevacizumab-IRDye800CW accumulates more in sinonasal inverted papilloma than in normal sinonasal mucosa.

Study design: The current study is a non-randomized, non-blinded, prospective, single center, pilot dose-escalation study. A minimum of five and a maximum of eight patients with SNIP will be included. Five patients will be administered with 10 mg bevacizumab-IRDye800CW. An interim analysis is performed after inclusion of the first three patients to determine if a tumor-to-background ratio (TBR) of ≥2 is obtained by either intraoperative fluorescence in vivo measurements or by ex vivo back-table fluorescence imaging. If a TBR of ≥2 is found, inclusion is continued to five patients. If not, the dose is adjusted to 25 mg. Again, a similar interim analysis is performed after inclusion of the first three patients to determine the TBR.

Study population: All included patients will meet the in- and exclusion criteria and have a biopsy confirmed diagnosis of primary or recurrent sinonasal inverted papilloma and are scheduled to undergo surgical resection.

Patient related study procedures: Patients will - after written informed consent - receive an intravenous injection of the fluorescent tracer. The dose will be either 10 mg or 25 mg. Two to four days later, the peroperative fluorescence imaging and multidiameter single fiber reflectance and single fiber fluorescence (MDSFR/SFF) spectroscopy will be performed of the tumor and woundbed.

Main study parameters/endpoints are macroscopic fluorescent signal levels, tumor to background ratio (TBR) and tracer distribution observed by fluorescence imaging and quantification of the fluorescent signal observed by means of MDSFR/SFF spectroscopy. Results of fluorescence imaging and spectroscopy will be correlated with standard histopathological assessment (i.e. hematoxylin and eosin staining) and VEGF immunohistochemistry.

Burden: Time investment: Patients need to visit the UMCG two to four days before their planned surgery which will take approximately two hours. Extra procedures: 1) Intravenous administration of bevacizumab-IRDye800CW. 2)The estimated time for taking fluorescence images and MDSFR/SFF spectroscopy measurements is approximately 15 minutes, which will result in prolongation of general anesthesia with 15 minutes. 3) Prior to surgical resection, the surgeon takes biopsies of fluorescent and non-fluorescent areas, or areas of inverted papilloma and normal mucosal lining of sinonasal cavities involved as identified by the surgeon when intraoperative fluorescent signal is not detected. 4) Immediately after resection of the inverted papilloma, biopsies will be taken from areas in the wound bed showing high fluorescent signal.

Risks: risks to study participants are mainly related to the, already present, risks of the surgical procedure and to the administration of the tracer in increasing dosages. A data safety monitoring board (DSMB) will not be installed as in more than two hundred patients receiving bevacizumab-IRDye800CW, no (serious) adverse events were observed.

Benefit: Patients will have no benefit from this study directly. Surgery will be planned as usual. During surgery, no decisions will be made based on the fluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of SNIP and scheduled to undergo surgical resection;
* Age ≥ 18 years;
* Written informed consent;
* Mentally competent person that is able and willing to comply with study procedures.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Concurrent uncontrolled medical conditions;
* Received an investigational drug within 30 days prior to the dose of bevacizumab-IRDye800CW;
* Tumors at sites of which the surgeon would assess that in vivo imaging would not be feasible;
* History of myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease or unstable angina within 6 months prior to enrollment;
* Inadequately controlled hypertension with or without current antihypertensive medications;
* History of infusion reactions to bevacizumab or other monoclonal antibody therapies;
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for women of childbearing potential. Woman of childbearing potential are premenopausal women with intact reproductive organs and women less than two years after menopause;
* Lab values that in the opinion of the primary surgeon would prevent surgical resection;
* Life expectancy < 12 weeks;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-to-background ratio of mean fluorescence intensity | Up to day 4

SECONDARY OUTCOMES:
Histopathologic assessment (H&E staining) of surgical specimen | Approximately two weeks
  Fluorescence signal will be correlated to histology of tissue (inverted papilloma, inflammation, malignant tumor, healthy tissue).
VEGF immunohistochemistry of surgical specimen | Approximately two weeks
  VEGF immunohistochemistry to correlate fluorescence signal with VEGF quantities

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vonk J, Voskuil FJ, de Wit JG, Heeman WT, Nagengast WB, van Dam GM, Feijen RA, Korsten-Meijer A, van der Vegt B, Witjes M. Fluorescence grid analysis for the evaluation of piecemeal surgery in sinonasal inverted papilloma: a proof-of-concept study. Eur J Nucl Med Mol Imaging. 2022 Apr;49(5):1640-1649. doi: 10.1007/s00259-021-05567-x. Epub 2021 Nov 5. PMID 34738141